CLINICAL TRIAL: NCT02426892
Title: Phase II Trial of Nivolumab and HPV-16 Vaccination in Patients With HPV-16-Positive Incurable Solid Tumors
Brief Title: Nivolumab and HPV-16 Vaccination in Patients With HPV-16 Positive Incurable Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: ISA Pharmaceuticals B.V. (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1047; NCI-2015-01004 (Registry Identifier: NCI CTRP Clinical Registry)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-12

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; HPV-16 Positive Incurable Solid Tumors; ISA101; HPV-16 vaccination; Nivolumab; BMS-936558; Opdivo
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ISA101 + Nivolumab (Experimental): HPV-16 vaccination (ISA 101) administered subcutaneously at 100 mcg for a total of 3 doses at 3 to 4 weeks intervals starting on Day 1.
  Nivolumab administered intravenously at 3 mg/kg every 2 weeks beginning on day 8 after the first vaccine dose.
  There are 3 weeks in Cycle 1 and 2 weeks in Cycles 2 and beyond.
  Interventions: Biological: ISA 101; Drug: Nivolumab

INTERVENTIONS:
Biological: ISA 101 — 100 mcg administered subcutaneously for a total of 3 doses at 3 to 4 weeks intervals starting on Day 1.
Drug: Nivolumab — 3 mg/kg administered by vein every 2 weeks beginning on Day 8 after the first vaccine dose.
  Other Names: BMS-936558; Opdivo

SUMMARY:
The goal of this clinical research study is to learn if nivolumab combined with ISA101 can help to control cancer that has spread. The safety of the study drugs will also be studied.

This is an investigational study. ISA101 is not FDA approved or commercially available. It is currently being used for research purposes only. Nivolumab is FDA approved to treat certain types of melanoma in patients who no longer respond to other drugs. Combining ISA101 with nivolumab is investigational. The study doctor can explain how the study drugs are designed to work.

Up to 28 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

There are 3 weeks in Cycle 1 and 2 weeks in Cycles 2 and beyond.

If you are found to be eligible to take part in this study, you will receive ISA101 by injection on Day 1 of Cycles 1, 2, and 4. You will be closely watched for the first 3 hours after each dose in order to check for any allergic reactions. Each time, you will receive 2 injections. One may be in your arm and one in your leg.

You will receive nivolumab by vein over 60 minutes on Day 8 of Cycle 1 and Day 1 of Cycles 2 and beyond.

Study Visits:

On Days 1 and 8 of Cycle 1 and Day 1 of every cycle after that:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests.

On Day 1 of Cycle 1 and then 1 time a month after that, if you can become pregnant, blood (about 1 teaspoon) or urine will be collected for a pregnancy test.

At Week 11 and every 6 weeks after that, you will have a CT scan or MRI to check the status of the disease.

Additional Research Tests:

Blood (up to 20 teaspoons each time) will be drawn before you begin to receive the study treatment, before you receive ISA101 at Weeks 3 and 7, before you receive nivolumab at Weeks 9 and 11, then every 12 weeks after that. If the doctor thinks it is needed because of white blood cell recovery from stored cells, one of the every 12 week blood draws may be done earlier. These blood samples will be used for biomarker tests and tests of the immune system.

Length of Treatment:

You may take ISA101 for up to 3 doses. You may continue taking nivolumab for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if intolerable side effects occur, or if you are unable to follow study directions.

If the disease seems like it has gotten worse, you may decide to continue to receive nivolumab, if you are still eligible. It is possible the study drug may be working even though the tumor(s) got larger. However, there are risks of continuing to receive the study drug because the disease may actually be getting worse. This is described in the side effects section below.

Your participation on the study will be over after the follow-up.

Follow-up Visits:

At about 30 days and 70 days after the last study drug dose, and then as often as the doctor decides as needed, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 4 teaspoons) will be drawn for routine tests.

At about 30 days, 70 days, and every 6 weeks after that (if you stop the study drug[s] for reasons other than the disease getting worse), you will have a CT or MRI scan to check the status of the disease. If the disease gets worse, these scans will stop.

Every 3 months for up to 3 years after your last study drug dose, you will be asked how you are doing (either at a visit or by phone). The calls should last about 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent: a. Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care. b) Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
2. Target Population: a. Men and women >/= 18 years of age. b. Eastern Cooperative Oncology Group (ECOG) performance status of </= 1. c. Subjects with histologically- or cytologically-documented incurable Human Papillomavirus (HPV)-16 positive solid tumors including oropharyngeal squamous cell carcinoma (OPSCC), cervical, vulvar, vaginal, anal, penile cancer. Incurable HPV-16 solid tumors are defined as tumors which are not curable by salvage approaches including resection and/or re-irradiation. HPV-16 serotype will be assessed by Cervista assay.
3. Target Population: Subjects can be treatment naïve for metastatic or incurable locally advanced HPV-16 positive solid tumors or can have one prior line of treatment.Patients are eligible upon progression after definitive local treatment (usually concurrent chemoradiation) if they are not candidates for salvage surgery or re-irradiation. Patients are also eligible after progression on first line chemotherapy for recurrent disease.
4. Target Population: d. Subjects must have measurable disease by CT or MRI per RECIST 1.1 criteria; Radiographic Tumor Assessment performed within 28 days of study inclusion. e. Target lesions may be located in a previously irradiated field if there is documented (radiographic) disease progression in that site. f. Subject entering the study will need to consent for mandatory biopsy at study entrance and as an optional procedure at week 11 and at progression for biomarker evaluation. Biopsy should be excisional, incisional or core needle. Fine needle aspiration is insufficient. g. Prior radiotherapy or radiosurgery must have been completed at least 2 weeks prior to start.
5. Target Population: h. All baseline laboratory requirements will be assessed and should be obtained within -14 days of study registration. Screening laboratory values must meet the following criteria: i) WBCs >/= 2000/uL; ii) Neutrophils >/= 1500/uL; iii) Platelets >/= 100 x 10^3/uL; iv) Hemoglobin >/= 9.0 g/dL; v) Serum creatinine of </= 1.5 X ULN or creatinine clearance > 40 mL/minute (using Cockcroft/Gault formula). Female CrCl= (140- age in years) x weight in kg x 0.85 72 x serum creatinine in mg/ dL. Male CrCl= (140- age in years) x weight in kg x 1.00 72 x serum creatinine in mg/ dL; vi) AST </= 1.5X ULN; vii) ALT </= 1.5X ULN; viii) Total bilirubin </= ULN (except subjects with Gilbert Syndrome who must have total bilirubin <3.0 mg/dl).
6. Age and Reproductive Status: a) Women of childbearing potential (WOCBP) must use method(s) of contraception for 30 days + 5 half-lives (60 days) of the study drugs. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. Highly effective birth control in this study is defined as a double barrier method. Examples include a condom (with spermicide) in combination with a diaphragm, cervical cap, or intrauterine device (IUD). The individual methods of contraception should be determined in consultation with the investigator. b) WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of investigational product.
7. Age and Reproductive Status: c) Women must not be breastfeeding. d) Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control for a period of 90 days plus the time required for the investigational drug to undergo 5 half-lives (60 days).

Exclusion Criteria:

1. Target Disease Exceptions: a. Subjects with active CNS metastases are excluded. Subjects are eligible if CNS metastases are adequately treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrollment. In addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of </= 10 mg daily prednisone (or equivalent) for 2 weeks. b. Subjects with carcinomatous meningitis.
2. Medical History and Concurrent Diseases: a. Subjects with active, known or suspected systemic autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll. b. Subjects with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of start. Inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease.
3. Medical History and Concurrent Diseases: c. Prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways). d. Subjects with a history of interstitial lung disease. e. Other active malignancy requiring concurrent intervention. f. Subjects with previous malignancies (except non-melanoma skin cancers, and the following in situ cancers: bladder, gastric, colon, endometrial, cervical/dysplasia, melanoma, or breast) are excluded unless a complete remission was achieved at least 2 years prior to study entry AND no additional therapy is required during the study period.
4. Medical History and Concurrent Diseases: g. Subjects with toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue that have not resolved to grade 1 (NCI CTCAE version 4) or baseline before administration of study drug. h. Subjects who have not recovered from the effects of major surgery or significant traumatic injury at least 14 days before the first dose of study treatment. i. Treatment with any investigational agent within 28 days of first administration of study treatment.
5. Physical and Laboratory Test Findings: a) Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS). b) Positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection.
6. Allergies and Adverse Drug Reaction: a) History of severe hypersensitivity reactions to other monoclonal antibodies. b) History of allergy or intolerance (unacceptable adverse event) to study drugs components.
7. Sex and Reproductive Status: a) WOCBP who are pregnant or breastfeeding. b) Women with a positive pregnancy test at enrollment or prior to administration of study medication
8. Prohibited Treatments and/or Restricted Therapies: a) Ongoing or planned administration of anti-cancer therapies other than those specified in this study. b) Use of corticosteroids or other immunosuppressive medications as per Exclusion Criteria 2b.
9. Other Exclusion Criteria: a) Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results. b) Prisoners or subjects who are involuntarily incarcerated. c) Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie S. Glisson, MD, BS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Sousa LG, Rajapakshe K, Rodriguez Canales J, Chin RL, Feng L, Wang Q, Barrese TZ, Massarelli E, William W, Johnson FM, Ferrarotto R, Wistuba I, Coarfa C, Lee J, Wang J, Melief CJM, Curran MA, Glisson BS. ISA101 and nivolumab for HPV-16+ cancer: updated clinical efficacy and immune correlates of response. J Immunother Cancer. 2022 Feb;10(2):e004232. doi: 10.1136/jitc-2021-004232. PMID 35193933
- [Derived] Massarelli E, William W, Johnson F, Kies M, Ferrarotto R, Guo M, Feng L, Lee JJ, Tran H, Kim YU, Haymaker C, Bernatchez C, Curran M, Zecchini Barrese T, Rodriguez Canales J, Wistuba I, Li L, Wang J, van der Burg SH, Melief CJ, Glisson B. Combining Immune Checkpoint Blockade and Tumor-Specific Vaccine for Patients With Incurable Human Papillomavirus 16-Related Cancer: A Phase 2 Clinical Trial. JAMA Oncol. 2019 Jan 1;5(1):67-73. doi: 10.1001/jamaoncol.2018.4051. PMID 30267032
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 participants were registered, 9 participants screen fail (not treated, not eligible or inevaluable)
Groups:
- ISA101 Vaccine and Nivolumab: Treatment with the ISA101 vaccine on days 1, 22 and 50. Nivolumab treatment IV starting day 8 of Cycle 1 and HPV-16 vaccination (ISA 101) administered subcutaneously at 100 mcg for a total of 3 doses at 3 to 4 weeks intervals starting on Day 1.
  Nivolumab administered intravenously at 3 mg/kg beginning on cycle 1 day 8 after the first vaccine dose and every two weeks there after until progression.
Period: Overall Study
Arm/Group | ISA101 Vaccine and Nivolumab
Started | 24
Completed | 4
Not Completed | 20
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 17
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All participants that signed the consent.
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 25
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response Rate (ORR)
Description: ORR defined as sum of subjects with a complete response (CR) and partial response (PR) divided by number of evaluable subjects at 11 weeks from start of treatment. RECIST 1.1 criteria used for assessment. CR is defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the time of the first protocol-specific intervention, every 6 weeks until progression, death, withdrawal of consent or study completion, an average of 4.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 24
Participants
  Complete Response (CR) | 2
  Partial Response (PR) | 6

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: PFS is defined as the time from first day of treatment to the date of the first documented tumor progression or death due to any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST V1.1). RECIST V1.1 defines progression as at least a 20% increase in the sum of diameters of target lesions, and the sum must also demonstrate an absolute increase of at least 5 mm. Additionally, the appearance of one or more new lesions is also considered progression. Progression Free survival will be summarized using the method of Kaplan and Meier and Cox proportional hazards model.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 24
months | 2.66 [2.5 to 9.44]

3. Secondary Outcome: Progression Free Survival (PFS) Rates at 2 and 3 Years
Description: as for outcome 2
Time Frame: From the time of the first protocol-specific intervention, every 6 weeks until progression, death, withdrawal of consent or study completion, an average of 3 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 24
months
  2 Years | 12.5 [4.3 to 36]
  3 Years | 12.5 [4.3 to 36]

4. Secondary Outcome: Median Overall Survival
Description: OS is defined as the time from treatment to the date of death, whichever comes first. Overall survival will be summarized using the method of Kaplan and Meier) and Cox proportional hazards model.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 24
months | 15.3 [10.6 to 27.2]

5. Secondary Outcome: Overall Survival (OS) Rates at 2 and 3 Years
Description: OS is defined as the time from treatment to the date of death. Overall survival will be summarized using the method of Kaplan and Meier) and Cox proportional hazards model.
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 24
months
  2 Years | 33 [18.9 to 58.7]
  3 Years | 12.5 [4.3 to 36]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: The safety and tolerability which will be measured by the incidence of adverse events, serious adverse events, deaths, and laboratory abnormalities. Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a subject or clinical investigation subject administered an investigational (medicinal) product and that does not necessarily have a causal relationship with this treatment. Laboratory abnormalities are Any laboratory test result that is clinically significant or meets the definition of an SAE, laboratory abnormality that required the subject to have study drug discontinued or interrupted, laboratory abnormality that required the subject to receive specific corrective therapy. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: at baseline, and continuously throughout the study at the beginning of each subsequent cycle, up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | ISA101 Vaccine and Nivolumab
Number analyzed (Participants) | 24
Participants
  Adverse Events | 23
  Serious Adverse Events | 11
  Death | 20
  Laboratory Abnormalities | 3

ADVERSE EVENTS:
Time Frame: Deaths, Serious Adverse Events and Other (Not Including Serious) Adverse events will be captured from the time of the first protocol-specific intervention, until 30 days after the last dose of drug, unless the participant withdraws consent, through study completion an average of 3 years.
Description: Number of participants affected 20, Number of Participants at Risk 24. 18 Patients affected died due to disease progression and all died greater than 30 days after last treatment on study. One died before starting treatment and one died at cycle 2 day 1 treatment, and both due to disease progression.
Arm/Group | ISA101 Vaccine and Nivolumab
All-Cause Mortality (participants affected / at risk) | 20/24
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISA101 Vaccine and Nivolumab (N=24)
Acute kidney injury (Renal and urinary disorders) | 1 (1) — (MedDRA v12.0,10069339)
lanine aminotransferase increased (Investigations) | 1 (1) — (MedDRA v12.0,10001551)
Anemia (Blood and lymphatic system disorders) | 1 (1) — (MedDRA v12.0,10002272)
Aspartate aminotransferase increased (Investigations) | 1 (1) — (MedDRA v12.0,10003481)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — (MedDRA v12.0,10003504)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) — (MedDRA v12.0,10010000)
Dysphagia (Gastrointestinal disorders) | 1 (1) — (MedDRA v12.0,10013950)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — (MedDRA v12.0,10013963)
Gastroparesis (Gastrointestinal disorders) | 1 (1) — (MedDRA v12.0,10018043)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — (MedDRA v12.0,10021881)
Lung infection (Infections and infestations) | 1 (1) — (MedDRA v12.0,10061229)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — (MedDRA v12.0,10028836)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) — (MedDRA v12.0,10030980)
Pancreatitis (Gastrointestinal disorders) | 1 (1) — (MedDRA v12.0,10033645)
Soft tissue infection (Infections and infestations) | 1 (1) — (MedDRA v12.0,10062255)
Syncope (Nervous system disorders) | 1 (1) — (MedDRA v12.0,10042772)
Thromboembolic event (Vascular disorders) | 1 (1) — (MedDRA v12.0,10043565)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — (MedDRA v12.0,10038738)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISA101 Vaccine and Nivolumab (N=24)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6)
Alkaline phosphatase increased (Investigations) | 6 (8)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 17 (44)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (10)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood and lymphatic system disorders - (bilirubin increased), specify (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 7 (9)
Blurred vision (Eye disorders) | 3 (3)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Chills (General disorders) | 6 (7)
Cholesterol high (Investigations) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16)
Creatinine increased (Investigations) | 3 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Depression (Psychiatric disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 7 (10)
Dizziness (Nervous system disorders) | 6 (7)
Dry mouth (Gastrointestinal disorders) | 8 (8)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 10 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (16)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema face (General disorders) | 5 (5)
Edema limbs (General disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eye disorders - (Other), specify (Eye disorders) | 2 (2)
Eye infection (Infections and infestations) | 1 (1)
Facial pain (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 19 (25)
Fever (General disorders) | 9 (14)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Flu like symptoms (General disorders) | 3 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
General disorders and administration site conditions - (diabetes type 2), specify (General disorders) | 1 (1)
General disorders and administration site conditions - (sensory neuropathy), specify (General disorders) | 1 (1)
General disorders and administration site conditions - (numbness), specify (General disorders) | 1 (1)
General disorders and administration site conditions - (Other), specify (General disorders) | 1 (1)
General disorders and administration site conditions - (left maxillary), specify (General disorders) | 1 (1)
General disorders and administration site conditions - (right parotitis was given anitbiotic), speci (General disorders) | 1 (1)
General disorders and administration site conditions - (possible related to nivolumab), specify - 10 (General disorders) | 1 (1)
Generalized muscle weakness - 10062572 / CTCAE4.03 (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 8 (9)
Hearing impaired (Ear and labyrinth disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hot flashes (Vascular disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 7 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (17)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3)
Hypoparathyroidism (Endocrine disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Hypothyroidism (Endocrine disorders) | 7 (9)
Infections and infestations - (possibly related to nivolumab MRSA and pneumonia), specify (Infections and infestations) | 1 (1)
Infections and infestations - (Cellulitis), specify (Infections and infestations) | 1 (1)
Infections and infestations - (Other), specify (Infections and infestations) | 1 (1)
Injection site reaction (General disorders) | 2 (2)
INR increased (Investigations) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5)
Investigations - (RELATED TO NIVO. INCREASE NEUTOROPHILE COUNT), specify (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (2)
Lung infection (Infections and infestations) | 1 (2)
Lymphedema (Vascular disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 8 (8)
Memory impairment (Nervous system disorders) | 1 (1)
Metabolism and nutrition disorders - (Possible related to Nivo), specify (Metabolism and nutrition disorders) | 1 (2)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Specify (not related to nivolumab) (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (22)
Neck edema (General disorders) | 1 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 1 (3)
Oral pain (Gastrointestinal disorders) | 2 (3)
Otitis media (Infections and infestations) | 1 (1)
Pain (General disorders) | 13 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Renal and urinary disorders - (nocturia), specify (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - (unlikely related to Nivo), specify (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - (Other), specify (Renal and urinary disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - (right vocal cord paralysis), specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - (secretions in the larynx/hypopharynx), specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scleral disorder (Eye disorders) | 1 (1)
Serum amylase increased (Investigations) | 1 (4)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - (shingles), specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - (lump at vaccine injection site related to vaccine), specif (Skin and subcutaneous tissue disorders) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 4 (5)
Skin infection (Infections and infestations) | 1 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (10)
Watering eyes (Eye disorders) | 1 (1)
Weight loss (Investigations) | 7 (7)
White blood cell decreased (Investigations) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT02426892/Prot_SAP_000.pdf